CLINICAL TRIAL: NCT02632773
Title: The Role of Parent Phenotype in Parent-Mediated Language Interventions for Autism
Brief Title: Parent Language Intervention for Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Megan Roberts, Jane Steiner Hoffman and Michael Hoffman Assistant Professor of Communication Sciences and Disorders, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01DC014709-01 (NIH); 1R01DC014709-01 (NIH)
Record Dates: First submitted 2015-12-08; First posted 2015-12-17 (Estimated); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Autism
Keywords: Language Intervention; Parent-Mediated Intervention
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Parent Learning Style 1 (Experimental): Mothers with Learning Style 2 will be randomly assigned to either the responsive intervention or directive intervention group.
  Interventions: Behavioral: Responsive Intervention
- Parent Learning Style 2 (Experimental): Mothers with Learning Style 2 will be randomly assigned to either the responsive intervention or directive intervention group.
  Interventions: Behavioral: Responsive Intervention
- Learning Style 1 (Parent) (Other): Mothers with Learning Style 2 will be randomly assigned to either the responsive intervention or directive intervention group.
  Interventions: Behavioral: Directive Intervention
- Learning Style 2 (Parent) (Other): Mothers with Learning Style 2 will be randomly assigned to either the responsive intervention or directive intervention group.
  Interventions: Behavioral: Directive Intervention

INTERVENTIONS:
Behavioral: Responsive Intervention — Mothers assigned to the responsive experimental condition will learn how to talk about what is in their child's focus of attention and to respond to all child communicative attempts by either: (a) assigning a presumed meaning to preverbal communication or vocalizations or (b) by repeating the child's verbal communication and adding words.
  Arms: Parent Learning Style 1; Parent Learning Style 2
Behavioral: Directive Intervention — Mothers assigned to the directive experimental condition will learn how to: (a) set up a prompting trial through management of toys or by responding to a child request, (b) recruit the child's attention, (c) provide a discriminative stimulus (cue), (d) wait for the child's response for 5 seconds, (e) reinforce the child for correct production of the target or provide additional prompts after incorrect productions. Parents will perform one prompting trial per minute for a total of 20 trials per parent session.
  Arms: Learning Style 1 (Parent); Learning Style 2 (Parent)

SUMMARY:
Improving social communication outcomes for children with autism spectrum disorders (ASD) has important public health implications. The proposed research is a randomized controlled trial of 108 children with ASD that examines how specific parent characteristics influence outcomes of two different parent-mediated language interventions. Evaluating effective language intervention strategies for children with ASD supports NIDCD's mission of behavioral research aimed to remediate the disordered process of language development in children with ASD.

DETAILED DESCRIPTION:
High dosage of early intervention is critical to language skill development in young children with autism spectrum disorders (ASD) and including parents is a cost-effective approach to maximize intervention dosage. However, parent-mediated interventions have inconsistent effects on parent and child outcomes. This variability is likely because parents do not have the same training as clinicians and little effort has been spent examining parent characteristics that may influence their ability to implement different types of intervention strategies. Given the known cognitive, personality and language features present among many parents of children with ASD, examining the relationship between learning styles in parents and their implementation of different parent-mediated intervention strategies is an important first step in identifying potential sources of variability in parent-mediated intervention outcomes. The objective of the proposed study is to examine how parent learning style influences parent use of language intervention strategies and subsequent child language skills. The central hypothesis is that the parent learning style will be associated with: (a) differential use of language intervention strategies and (b) child language skills. The specific aims include determining the extent to which: (a) parent learning style and type of parent-mediated intervention are associated with mother use of language intervention strategies and subsequent child language skills, (b) parent learning style moderates the relationship between intervention type and mother use of language intervention strategies, and (c) parent learning style is associated with their use of language intervention strategies and their children's language skills. The proposed study will enroll 108 children with ASD between 24 and 36 months of age and their mothers. Mother-child dyads will be randomly assigned to one of two parent-mediated intervention strategies that are contrasted in their theoretical approach (responsive-developmental, directive-behavioral). Mother-child dyads will be assessed before randomization (pre-test), after intervention (post-test) and 3 months after the end of intervention to monitor maintenance. Children in both groups will receive 8 weekly intervention sessions at home using the same experimental procedures. The proposed research is significant because it will be the first examination of the impact of parent learning style on both parent and child outcomes of two different parent-mediated intervention strategies (directive, responsive). Understanding the effects of parent learning style on parent use of intervention strategies and subsequent child language skills is a key step in customizing parent-mediated interventions based on parent characteristics. The long-term positive effect of the proposed research is to improve language outcomes of interventions for children with autism by tailoring parent-mediated interventions that capitalize on parental strengths.

ELIGIBILITY:
Inclusion Criteria:

Child inclusion criteria include:

* diagnosis of ASD based on ADOS
* chronological age of less than 48 months
* a parent who is willing to learn intervention strategies
* English as the primary language spoken in the home

Parent Inclusion Criteria Include:

- Mother

Exclusion Criteria:

* Children or parents with additional impairments (e.g., blindness, deafness, genetic syndromes) will be excluded from the study.
* Fathers or caregivers other than the child's Mother will be excluded from the study.

Ages: 18 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Parent Use of Language Support Strategies (Mother-child interaction) | Two months after the start of the study
  Mother use of intervention strategies will be measured by transcribing and coding mother behaviors during parent-child interactions.

SECONDARY OUTCOMES:
Expressive vocabulary of the child as measured by transcribing and coding a 20 minute video of a therapist-child interaction in the clinic with a standard set of age-appropriate toys. | Two months after the start of the study
  20 minute video of a therapist-child interaction in the clinic with a standard set of age-appropriate toys.
MacArthur-Bates Communicative Development Inventory (MCDI) (Child) | Two months after the start of the study
  Parent report of child's expressive vocabulary and prelinguistic communication skills

CONTACTS AND LOCATIONS:
Overall Officials: Megan Y Roberts, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Sharing baseline data with the National Database for Autism Research (NDAR) semi-annually.

REFERENCES:
- [Background] Roberts MY, Kaiser AP. Early intervention for toddlers with language delays: a randomized controlled trial. Pediatrics. 2015 Apr;135(4):686-93. doi: 10.1542/peds.2014-2134. Epub 2015 Mar 2. PMID 25733749
- [Derived] Fipp-Rosenfield HL, Levy RS, Grauzer JM, Kaat A, Roberts MY. Autistic Children's Irritability During Social Communication Assessments. Am J Speech Lang Pathol. 2024 Jan 3;33(1):369-377. doi: 10.1044/2023_AJSLP-23-00216. Epub 2023 Nov 27. PMID 38010261